CLINICAL TRIAL: NCT03249311
Title: Effectiveness of the Norepinephrine and Serotonin Reuptake Inhibitor Levomilnacipran in Healthy Males
Brief Title: Levomilnacipran in Healthy Males
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Ottawa (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Pierre Blier, Endowed Research Chair and Director of Mood Disorders Research Unit, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: REB2017004
Record Dates: First submitted 2017-07-20; First posted 2017-08-15 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: None (i.e. Healthy Volunteers)
Keywords: Levomilnacipran; Antidepressant; Ottawa; Selective Norepinephrine Reuptake Inhibitor; Healthy males; Tyramine response; Serotonin; Norepinephrine
MeSH Terms: interventions — Levomilnacipran; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Levomilnacipran (Experimental): Participants will be randomly assigned to receive levomilnacipran, duloxetine, or placebo
  Interventions: Drug: Levomilnacipran
- Duloxetine (Cymbalta) (Active Comparator): Participants will be randomly assigned to receive levomilnacipran, duloxetine, or placebo
  Interventions: Drug: Duloxetine
- Levomilnacipran Placebo-matched capsules (Placebo Comparator): Participants will be randomly assigned to receive levomilnacipran, duloxetine, or placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Levomilnacipran — Escalating doses of 40 to 120mg/day every 7 days (+/- 1 day) throughout a 20-26 day period.
  Other Names: Fetzima
  Arms: Levomilnacipran
Drug: Duloxetine — Escalating doses of 40 to 120mg/day every 7 days (+/- 1 day) throughout a 20-26 day period.
  Other Names: Cymbalta
  Arms: Duloxetine (Cymbalta)
Drug: Placebos — Escalating doses of 40 to 120mg/day every 7 days (+/- 1 day) throughout a 20-26 day period.
  Arms: Levomilnacipran Placebo-matched capsules

SUMMARY:
Levomilnacipran is an antidepressant currently approved in Canada to treat Major Depressive Disorder (MDD). Thirty-six healthy male participants will receive escalating doses of levomilnacipran, duloxetine, or placebo every 7 days (+/- 1 day) throughout a 20 - 28 day period. After each dose escalation study participants will be asked to come to the clinic to conduct the necessary tests - these will include tyramine pressor tests as well as blood draws. The results of this study will allow the investigators to determine the dose(s) of levomilnacipran at which reuptake inhibition of norepinephrine and serotonin (chemicals utilized by nerve cells to transmit information to other cells) is achieved.

DETAILED DESCRIPTION:
Levomilnacipran (Fetzima) is the active enantiomer of milnacipran (Ixel, Savella) for norepinephrine (NE) and serotonin (5-hydroxytryptamine, 5-HT) reuptake. It has an approximate eight-fold greater affinity for the human NE transporter than for the 5-HT transporter. This signifies that the NE transporter may be engaged to a much greater degree than the 5-HT transporter at various doses, especially at lower regimens. As such, levomilnacipran represents the mirror antidepressant medication of venlafaxine and duloxetine since at their minimal effective doses, these medications are selective inhibitors of 5-HT reuptake and it is not until daily regimens are doubled or tripled that the NE transporter gets engaged.

Levomilnacipran is effective clinically in patients with major depressive disorder (MDD) at doses ranging between 40 and 120 mg/day. Given this wide effective dose range, it appears essential to determine the in vivo potency of levomilnacipran and the dose at which it starts inhibiting 5-HT in relation to NE reuptake in humans.

The current investigators have studied the NE reuptake blocking properties of antidepressants in both healthy volunteers and patients with depression using tyramine pressor tests. This peripheral model of adrenergic function involves administration of repeated intravenous injections of tyramine and measurement of transient increases in systolic blood pressure (SBP) that occur after a tyramine load. This approach has led to dose-dependent SBP increases that are reliably reproduced one week apart in healthy volunteers who received placebo which supports the use of the tyramine pressor test to assess the functional capacity of different medication regimens to inhibit NE reuptake at steady state levels. Serotonin reuptake has been extensively studied in human participants using the blood platelet model. In this assay, whole blood 5-HT and/or platelet content is determined before and after giving reuptake inhibitors. Since the 5-HT transporter is similar on 5-HT neurons in the brain and on platelets, the degree of 5-HT depletion in the blood can be used as a measure of 5-HT reuptake blockade in the brain. Together, these experimental approaches will identify the potency of levomilnacipran for NE and 5-HT reuptake inhibition.

The purpose of this study is to determine the potency of levomilnacipran required to inhibit NE and 5-HT reuptake in healthy male participants across the effective dose range of the medication (40-120 mg/day).

Participants Healthy male participants will receive escalating doses of levomilnacipran, duloxetine, or placebo every 4-7 days throughout a 14-23 day period. The tyramine pressor procedure will be used to identify the dose at which these medications inhibit norepinephrine reuptake. Serotonin reuptake inhibition will be estimated from whole blood serotonin concentrations. Tyramine testing and blood draws will occur at baseline (prior to medication administration) and 4 days after each dose escalation.

Participants will be assigned to one of 3 groups: levomilnacipran, duloxetine or placebo. The duration of study treatment for participants in the first 2 groups will range from 22-32 days. These participants will receive escalating doses of levomilnacipran or duloxetine over a period of 14-23 days followed by down-titrated doses over the next 8 days. The investigators will offer a flexible interval for dose escalation in participants receiving levomilnacipran and duloxetine to minimize side effects, improve tolerability, and maximize subject retention. Participants in the placebo group will receive the levomilnacipran-matched placebo capsule for 14 days.

Specific aim The objective of this study is to assess the norepinephrine and serotonin reuptake inhibition capacities of levomilnacipran using the tyramine pressor procedure and blood platelet model respectively. Two control groups will be included to demonstrate the validity of the two experimental approaches, an active comparator group, and a placebo group. Therefore, there will be three treatment arms: 1) 12 participants will be administered escalating doses of levomilnacipran, 2) 12 participants will be administered escalating doses of duloxetine, and 3) 12 participants will receive levomilnacipran placebo-match capsules. Duloxetine will be used as an active comparator as it is an established 5-HT reuptake inhibitor and a potentially effective NE reuptake inhibitor.

Assessments to be Performed Pharmacodynamic and safety evaluations: At each visit, a catheter will be placed in the subject's antecubital vein. The participant will lie down and remain supine until his pulse is determined to be stable (+/- approximately 5 bpm) over two consecutive measurements made a minimum of 10 minutes apart. The subject's heart rate and blood pressure will be recorded from the arm contralateral to the catheter. Blood samples will be drawn from the catheter while the participant remains supine. The participant's heart rate and blood pressure will again be recorded from the arm contralateral to the catheter.

Plasma drug levels: Plasma concentrations of levomilnacipran and duloxetine will be determined from supine blood samples after each dose change to ensure that potentially aberrant results are not due to poor medication compliance.

Whole blood serotonin assay: Whole blood 5-HT concentrations will be determined from supine blood samples collected at regular visits.

Evaluation of tyramine pressor response: After the supine blood samples are drawn, the tyramine infusion procedure will proceed as follows: 1) The participant will be connected to the cardiac monitor apparatus, which automatically monitors blood pressure and heart rate. 2) The participant will lie down and remain supine until his pulse is determined to be stable over two consecutive measurements made a minimum of 10 minutes apart. 3) A first small dose of tyramine (0.5 mg) will be administered intravenously to rule out the presence of pheochromocytoma. Pheochromocytoma is a small neuroendocrine tumour which can cause elevated secretion of catecholamines leading to raised blood pressure, palpitations and headaches. This condition would not be detected through physical exam or laboratory tests. This dose is not expected to produce any significant change in the cardiovascular parameters measured. Ten minutes after the participant receives the 0.5 mg tyramine dose, the effects of two fixed doses of intravenous tyramine on systolic blood pressure will be assessed. First, a 4 mg dose of tyramine will be administered. Five minutes after the subject's blood pressure returns to normal, a 6 mg dose will be administered. 4) Heart rate, systolic and diastolic blood pressure will be recorded every 2 minutes for at least 10 minutes after the injection, or 5 minutes after the return of baseline blood pressure and heart rate, whichever is longer.

Safety/Monitoring procedures: A physician and research nurse coordinator will be present during the entire tyramine procedure, and participants will remain on the unit for a further 15 min after all Tyramine Pressor Test procedures have completed for monitoring. There is access to an automated external defibrillator (AED), and a crash cart with supporting staff in case of emergency.

ELIGIBILITY:
Inclusion Criteria:

* Male participants between 18 and 40 years-old
* Written informed consent signed by the participant

Exclusion Criteria:

* Lifetime personal history of diagnosis of major depressive disorder according to the DSM-V (American Psychiatric Association, 2013) using the Structured Clinical Interview for DSM-V Axis I Disorders, Research Version, Non-patient Edition (SCID-5-RV for DSM-V; First et al., 2015)
* A history of suicidal ideation and behaviour, including self-harm and/or harm to others.
* A history of substance abuse and/or dependence.
* A positive drug screen for illicit drugs
* Substantial alcohol use
* Current use of Monoamine Oxidase Inhibitors (MAOIs), including the antibiotic linezolid and the thiazine dye methylthioninium chloride (methylene blue)
* Current use of serotonin-precursors (such as L-tryptophan, oxitriptan)
* Current use of serotonergic drugs (triptans, certain tricyclic antidepressants, lithium, tramadol, St. John's Wort)
* Concomitant use of NSAIDS, ASA, and other anticoagulants.
* Current use of Thioridazine
* Current use of CYP1A2 Inhibitors
* Current use of Triptans (5HT1 Agonists)
* Blood pressure greater than 140/90 and/or a pulse rate greater than 90 bpm
* Recent history of myocardial infarction, cerebrovascular accident, cardiac arrhythmias, or unstable heart disease.
* Evidence of significant physical illness contraindicating the use of levomilnacipran and duloxetine found on the physical exam or in the laboratory data obtained during the first week of the study
* Current use of medication that may affect voiding (ie- anticholinergics)
* History of obstructive urinary disorders and dysuria, prostatic hypertrophy, prostatitis, and other lower urinary tract obstructive disorders.
* History of Stevens-Johnson Syndrome and Erythema multiforme.
* Diabetes Type I and II
* Fructose intolerance, glucose-galactose malabsorption or sucrose-isomaltase insufficiency.
* Hepatic Impairment
* Uncontrolled narrow-angle glaucoma
* Severe renal impairment
* History of seizure disorder
* Anatomically narrow ocular angles.
* Osteoporosis or major risk for bone fractures.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary End Point | 24 months
  The degree of norepinephrine reuptake in response to the increasing levels of the study medication will be assessed and compared between three treatment groups.

SECONDARY OUTCOMES:
Secondary End Points | 24 months
  The degree of serotonin reuptake in response to the increasing levels of the study medication will be assessed and compared between three treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Blier, MD, Principal Investigator — The Royal's Institute of Mental Health Research
Locations (1):
- Institute of Mental Health Research, Royal Ottawa Mental Health Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asnis GM, Henderson MA. Levomilnacipran for the treatment of major depressive disorder: a review. Neuropsychiatr Dis Treat. 2015 Jan 9;11:125-35. doi: 10.2147/NDT.S54710. eCollection 2015. PMID 25657584
- [Background] Auclair AL, Martel JC, Assie MB, Bardin L, Heusler P, Cussac D, Marien M, Newman-Tancredi A, O'Connor JA, Depoortere R. Levomilnacipran (F2695), a norepinephrine-preferring SNRI: profile in vitro and in models of depression and anxiety. Neuropharmacology. 2013 Jul;70:338-47. doi: 10.1016/j.neuropharm.2013.02.024. Epub 2013 Mar 13. PMID 23499664
- [Background] Blier P, Saint-Andre E, Hebert C, de Montigny C, Lavoie N, Debonnel G. Effects of different doses of venlafaxine on serotonin and norepinephrine reuptake in healthy volunteers. Int J Neuropsychopharmacol. 2007 Feb;10(1):41-50. doi: 10.1017/S1461145705006395. Epub 2006 May 11. PMID 16690005
- [Background] Aldosary F, Norris S, Tremblay P, James JS, Ritchie JC, Blier P. Differential Potency of Venlafaxine, Paroxetine, and Atomoxetine to Inhibit Serotonin and Norepinephrine Reuptake in Patients With Major Depressive Disorder. Int J Neuropsychopharmacol. 2022 Apr 19;25(4):283-292. doi: 10.1093/ijnp/pyab086. PMID 34958348
- [Background] Debonnel G, Saint-Andre E, Hebert C, de Montigny C, Lavoie N, Blier P. Differential physiological effects of a low dose and high doses of venlafaxine in major depression. Int J Neuropsychopharmacol. 2007 Feb;10(1):51-61. doi: 10.1017/S1461145705006413. Epub 2006 May 11. PMID 16690006
- [Background] First, M.B., Williams, J.B.W., Karg, R.S., & Spitzer, R.L. (2015). Structured clinical interview for DSM-5-research version. Arlington: American Psychiatric Association.
- [Background] Gobbi G, Slater S, Boucher N, Debonnel G, Blier P. Neurochemical and psychotropic effects of bupropion in healthy male subjects. J Clin Psychopharmacol. 2003 Jun;23(3):233-9. doi: 10.1097/01.jcp.0000084023.22282.03. PMID 12826985
- [Background] Turcotte JE, Debonnel G, de Montigny C, Hebert C, Blier P. Assessment of the serotonin and norepinephrine reuptake blocking properties of duloxetine in healthy subjects. Neuropsychopharmacology. 2001 May;24(5):511-21. doi: 10.1016/S0893-133X(00)00220-7. PMID 11282251
- [Background] Vincent S, Bieck PR, Garland EM, Loghin C, Bymaster FP, Black BK, Gonzales C, Potter WZ, Robertson D. Clinical assessment of norepinephrine transporter blockade through biochemical and pharmacological profiles. Circulation. 2004 Jun 29;109(25):3202-7. doi: 10.1161/01.CIR.0000130847.18666.39. Epub 2004 Jun 7. PMID 15184278
- [Derived] Nikolitch K, Phillips JL, Daniels S, Blier P. Levomilnacipran, but Not Duloxetine, Inhibits Serotonin and Norepinephrine Reuptake Throughout Its Therapeutic Range. J Clin Psychiatry. 2025 Aug 25;86(3):25m15867. doi: 10.4088/JCP.25m15867. PMID 40875503